



Centre Number:

Study Number: 242203

Name of Researcher: Dr Deborah Antcliff

Participant Identification Number for this study:

## **CONSENT FORM**

## Title of the study: Developing an activity pacing framework for the management of chronic

| | iio oi iiio otaayi b | | Stage III: Feasibility study | |
|---|---|---|---|---|
| | | | Pic | ease initial box |
| 1. | | had the opportunity to cor | t dated 27.04.2018 (Version 2.1) for the nsider the information, ask questions and have | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | | |
| 3. | I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from The Pennine Acute Hospitals NHS Trust or from regulatory authorities, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | rom |
| 4. | I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. | | | |
| 5. | I agree to take part in | n the above study. | | |
| Name of Participant | | Date | Signature | |
| Name of Person taking consent | | Date | Signature | |